CLINICAL TRIAL: NCT02102906
Title: TMS and Attentional Bias in Functional Motor Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMS
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2014-12

CONDITIONS: Conversion Disorder
Keywords: Adult; Humans; Conversion disorder; Somatoform Disorders/therapy; Nervous System Disorders/therapy
MeSH Terms: conditions — Conversion Disorder; Somatoform Disorders; Nervous System Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMS treatment (Experimental): Patients will receive a single session of 20 single pulses of TMS to motor cortex contralateral to affected upper limb at 120% motor threshold, with verbal encouragement throughout. Half of the patients recruited will be randomised to a 3 month delay during which they will receive treatment as normal.
  Interventions: Procedure: Transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Transcranial magnetic stimulation — Single pulse TMS - 20 pulses at 120% motor threshold. Using the Magstim rapid 2 stimulator, which has a CE mark and will be used within the indications specified by the CE mark.

SUMMARY:
Functional motor disorders, also called motor conversion disorder, are common reasons for attendance at neurology outpatient clinics. Patients with functional motor disorders are more common than patients with multiple sclerosis and have similar levels of disability but more psychological morbidity.

There is limited evidence for effective treatments in functional motor disorders. A small number of studies of transcranial magnetic stimulation (TMS), a painless method of cortical stimulation, have reported improvement in functional weakness after this treatment including in patients with symptoms of several years duration. The Investigators intend to trial TMS in a group of 40 patients with functional motor disorder, randomising patients to immediate or delayed treatment and therefore comparing a single session of TMS with routine clinical care. The Investigators will also ask patients to undergo tests of attentional focus in a cognitive neuroscience laboratory - these experiments will be analysed separately from TMS trial data.

DETAILED DESCRIPTION:
A randomised non-blinded controlled study design will be used, with 3 months of treatment as usual as the control condition and a single session of TMS as the treatment condition.

40 patients with functional unilateral upper limb weakness will be recruited from neurology and neuropsychiatry clinics in Edinburgh and randomised to either immediate treatment or to 3 month delay during which they will receive routine clinical care. Randomisation will be performed using computerised random number generator by a person not involved with the study.

Patients randomised to delay will complete baseline measures of disability and motor function including SF36, modified Rankin score and study specific questionnaires, and will repeat these after 3 months. Patients undergoing immediate treatment will complete the same questionnaires immediately before and 3 months after treatment. All individuals receiving TMS treatment will undergo tests of grip strength and tapping frequency immediately before and after treatment.

The treatment and experiments involved will be as follows. Patients will attend the PPLS Cognitive Neuroscience Laboratory at George Square, University of Edinburgh for a single 2 hour session. During the first hour they will complete baseline symptom severity and disability questionnaires and will undertake a series of 3 experiments. Experiments involve participants sitting with their head on a chin-rest looking at either a computer screen or at lights projected onto their own hands, and for one experiment with a vibrating 'buzzer' taped to each hand. They will be asked to respond verbally in experiments which test their response to distracting attentional 'cues' either visual or vibrotactile. These experiments will take less than 1 hour. In anaylsis, performance will be compared between affected and unaffected sides (ie left hand and right hand), and will also be compared with performance of a group of 15 healthy control participants recruited from spouses or partners.

Patient participants will then receive treatment with 20 single pulses of TMS to the motor cortex at 120% motor threshold. These will cause visible and palpable 'jerks' of the affected limb. Between stimulations the researcher will offer verbal encouragement and ask the participant to move the affected limb if possible. Treatment will take less than 1 hour.

The primary outcome measures are patient-rated symptom severity and disability and simple statistical analysis will be used to compare outcome after 3 months of treatment as normal and 3 months after a single session of TMS treatment. Secondary outcome measures include grip strength and tapping frequency before and after treatment. Data will be analysed on an intention-to-treat basis. Data from attentional tests will be analysed separately.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis, by a consultant neurologist, of functional motor disorder
* functional unilateral upper limb weakness present for 50% or more of the time
* age 18-75
* ability to give informed consent

Exclusion Criteria:

* difficulties in understanding spoken or written English
* history of epileptic seizures (non-epileptic seizures will not be an exclusion criteria)
* alcohol dependence
* severe co-morbid physical or psychiatric disorder
* factitious disorder
* patients unable to receive TMS because of metal implants such as pacemakers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patient-rated disability | An average of 3 months after day of attendance for TMS treatment.
  SF36 score and Modified Rankin Score
Patient rated symptom severity | An average of 3 months after day of attendance for TMS treatment
  Assessed using a Likert scale.

SECONDARY OUTCOMES:
Grip strength | Between 10 minutes and one hour before TMS treatment, and between 10 minutes and 1 hour after TMS treatment.
Hand tapping frequency | Between 10 minutes and one hour before TMS treatment, and between 10 minutes and 1 hour after TMS treatment
Patient rated treatment discomfort | Between 10 minutes and 1 hour after TMS treatment.

OTHER OUTCOMES:
Attentional focus / distractibility | Tests performed during the 1-2 hours before treatment.
  A short series of neurocognitive experiments based on a modified Posner test will examine for differences in attentional focus between affected and unaffected limbs and will also compare performance with a group of healthy controls recruited from spouses.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Stone, MBChB PhD FRCP, Principal Investigator — NHS Lothian
Locations (2):
- United Kingdom (2):
  - Department of Clinical Neurosciences, Western General Hospital, Edinburgh, Scotland
  - Department of Psychology, University of Edinburgh, Edinburgh, Scotland

REFERENCES:
- [Derived] McWhirter L, Ludwig L, Carson A, McIntosh RD, Stone J. Transcranial magnetic stimulation as a treatment for functional (psychogenic) upper limb weakness. J Psychosom Res. 2016 Oct;89:102-6. doi: 10.1016/j.jpsychores.2016.08.010. Epub 2016 Aug 25. PMID 27663118